CLINICAL TRIAL: NCT06178549
Title: Feasibility and Effectiveness of HPV Self-Sampling for Cervical Cancer Screening Among Women Seeking Health Care At a Safety Net Hospital Emergency Room
Brief Title: Emergency Room HPV Self-Sampling Study (ACT NOW)
Acronym: ACT NOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Aaron Peter Thrift, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H-52653
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (single arm) (Experimental): Intervention arm to complete HPV self-sampling
  Interventions: Behavioral: HPV Self-Sampling

INTERVENTIONS:
Behavioral: HPV Self-Sampling — HPV self-sampling. Participants will be provided with education regarding cervical cancer prevention and Aptima kit and instructions for self-sampling. Patient navigators will assist participants with positive HPV test results to connect with healthcare providers for follow-up screening and care.

SUMMARY:
The goal of this study is to develop and evaluate an evidence-based public health intervention using HPV self-sampling approach in an opportunistic setting to increase cervical cancer screening among screening non-attendees, particularly those uninsured or underinsured, who use emergency services to access medical care. The proposed pilot study will examine the feasibility and efficacy of HPV self-sampling among women at a safety net hospital emergency room. Participant recruitment and self-sample will take place in the waiting rooms in the ER. All women sitting in the waiting room will serve as the source population for the study and will be approached and invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are women ages 25 years to 65 years, with a cervix, presenting in the waiting areas at the Ben Taub General Hospital Emergency Department

Exclusion Criteria:

* Women under 25 years or older than 65 years of age,
* self-reported current pregnancy,
* self-reported history of cervical cancer,
* past hysterectomy,
* had Pap Smear within past 3 years or HPV/Pap co-test within past 5 years.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
HPV self-sampling completion | 1 day
  Participation rate for self-sample HPV testing (percent of eligible women who complete self-sampling).

SECONDARY OUTCOMES:
HPV self-sampling acceptability | 1 day
  acceptability of self-sample HPV testing using the global acceptability score
Attendance for cervical cancer screening among HR-HPV positive women | 6 months
  Rate of attendance for cervical cancer screening among HR-HPV positive women (percent of HR-HPV positive participants who obtain a Pap test following self-sample HPV testing)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No